CLINICAL TRIAL: NCT04505475
Title: Oral Surgery in Patients Taking Direct Oral Anticoagulants and Vitamin K Antagonists
Brief Title: Oral Surgery in Patients Taking Direct Oral Anticoagulants
Acronym: OSDOA
Status: Completed | Type: Observational
Sponsor: University of Novi Sad (Other)
Responsible Party: Principal Investigator, Branislav Bajkin, Principal Investigator, University of Novi Sad
Other Study IDs: 01-11/45-2015 DCV
Record Dates: First submitted 2020-08-05; First posted 2020-08-10 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Anticoagulants and Bleeding Disorders; Surgery; Postoperative Hemorrhage; Dentoalveolar Haemorrhage
Keywords: oral anticoagulants; dabigatran; rivaroxaban; warfarin; oral surgery; hemorrhage
MeSH Terms: conditions — Hemostatic Disorders; Postoperative Hemorrhage; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Direct oral anticoagulants: Patients taking dabigatran, ravaroxaban or apixaban
  Interventions: Procedure: Oral surgical procedure followed by local hemostatic measures (insertion of gelatine sponge and wound suturing)
- Vitamin K antagonists: Patients taking acenocoumarol with therapeutic INR levels (2.0-3.5)
  Interventions: Procedure: Oral surgical procedure followed by local hemostatic measures (insertion of gelatine sponge and wound suturing)

INTERVENTIONS:
Procedure: Oral surgical procedure followed by local hemostatic measures (insertion of gelatine sponge and wound suturing) — single and multiple teeth extraction, surgical tooth extraction, third molar surgery, gingivectomy, soft-tissue biopsy

SUMMARY:
This study evaluates the incidence of postoperative bleeding after oral surgical procedures in patients taking direct oral anticoagulants and in patients taking vitamin K antagonists.

DETAILED DESCRIPTION:
Vitamin K antagonists (VKA) are widely used in long term prevention and treatment of thromboembolism. In the last few years direct oral anticoagulants (DOACs) are available for clinical use, mostly in prevention of stroke and systemic embolisms in patients with nonvalvular atrial fibrillation, and prevention and treatment of venous thrombosis. Numerous studies confirmed that minor oral surgical procedures in patients taking VKA with therapeutic (International Normalized Ratio) INR levels can be safely performed without therapy interruption if proper local haemostatic measures are applied. Similar recommendations were given for the dental treatment of patients taking DOACs, but there is a lack of clinical studies. The aim of this study is to assess the incidence of bleeding complications after oral surgery in patients who continue their DOACs or VKA medications.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients over 18 years
* Patients taking regularly direct anticoagulant therapy: dabigatran, rivaroxaban or apixaban (DOACs group)
* Patients taking regularly acenocoumarol with INR 2.0-3.5 on the day of the surgery (VKA group)
* Indication for oral surgical procedure
* Signed informed consent

Exclusion Criteria:

* Liver or renal disease
* Coagulopathy
* Pregnant or breastfeeding women
* Allergy to lidocaine
* Patients who stopped taking their anticoagulant medication
* Patients taking VKA with INR <2.0 or >3.5 on the day of the procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study includes patients taking direct oral anticoagulants (DOACs) and patients taking vitamin K antagonists (VKA) who require oral surgical procedure. The groups will be matched with respect to oral surgical procedure i.e. operative trauma.
Sampling Method: Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2015-05-25 (Actual); Primary Completion 2020-08-03 (Actual); Study Completion 2020-08-03 (Actual)

PRIMARY OUTCOMES:
Postoperative bleeding event | 7 days
  Bleeding that requires additional surgical procedure

CONTACTS AND LOCATIONS:
Overall Officials: Branislav Bajkin, PhD, Principal Investigator — University of Novi Sad, Faculty of Medicine
Locations (1):
- Dental Clinic of Vojvodina, Novi Sad, Vojvodina, Serbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bajkin BV, Tadic AJ, Komsic JJ, Vuckovic BA. Risk of dentoalveolar surgery postoperative bleeding in patients taking direct oral anticoagulants and vitamin K antagonists: A prospective observational study. J Craniomaxillofac Surg. 2024 Jun;52(6):772-777. doi: 10.1016/j.jcms.2024.03.035. Epub 2024 Apr 1. PMID 38580558